CLINICAL TRIAL: NCT03865706
Title: Prebiotic Inulin to Limit Antimicrobial-Resistant Infections During Critical Illness: A Phase II Clinical Trial
Brief Title: Inulin for Infections in the Intensive Care Unit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel Freedberg, MD, Assistant Professor of Medicine and Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAS2576; PR181960 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Antibiotic Resistant Infection; Nosocomial Infection; Pathogen Transmission; Nutrition Disorders; Critical Illness; Sepsis
Keywords: Microbiome; Antibiotic resistance; Intensive care unit; Sepsis; Nutrition; Pathogen colonization
MeSH Terms: conditions — Cross Infection; Nutrition Disorders; Critical Illness; Sepsis | interventions — Inulin; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: placebo-controlled trial with 1:1:1 enrollment into three arms: inulin 32 g/day, inulin 16 g/day, and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Inulin 32 g/day (Experimental): Critically ill adults who are receiving broad-spectrum antibiotics will also receive inulin oral suspension (16g twice daily) for a minimum of 7 days.
  Interventions: Drug: Inulin Oral Suspension; Drug: Broad-spectrum antibiotics
- Inulin 16 g/day (Experimental): Critically ill adults who are receiving broad-spectrum antibiotics will also receive inulin oral suspension (8g twice daily) for a minimum of 7 days.
  Interventions: Drug: Inulin Oral Suspension; Drug: Broad-spectrum antibiotics
- Placebo (Placebo Comparator): Critically ill adults who are receiving broad-spectrum antibiotics will also receive placebo oral suspension for a minimum of 7 days.
  Interventions: Drug: Placebo Oral Suspension; Drug: Broad-spectrum antibiotics

INTERVENTIONS:
Drug: Inulin Oral Suspension — Inulin powder, derived from chicory root and re-suspended in 250cc water Dosage will be either 8g twice a day or 16g twice a day - dissolved in 250cc sterile water, given oral or via enteric tube
  Other Names: Inulin
  Arms: Inulin 16 g/day; Inulin 32 g/day
Drug: Placebo Oral Suspension — 250cc sterile water alone, given twice daily a sweetener is added to the water to create identical flavor
  Other Names: Placebo
  Arms: Placebo
Drug: Broad-spectrum antibiotics — Standard of care treatment for infections
  Other Names: Antibiotics

SUMMARY:
Normal gut bacteria prevent colonization and subsequent infection with MDR organisms (MDROs) through competition for resources and other mechanisms. During critical illness, this function of the microbiome is lost and there are no current treatments to restore it. Preliminary data indicates that the prebiotic fiber inulin is safe and may alter the gastrointestinal microbiome to improve gut barrier function, decrease colonization with MDROs, and reduce downstream risk for intensive care unit (ICU)-acquired MDR infections. However, the impact of inulin during critical illness is unknown. This double-blind, randomized clinical trial will test inulin for the prevention of antibiotic resistant infections in the ICU.

The trial's specific aims are to determine (1) the feasibility, tolerability, and safety of inulin in the intensive care unit; (2) the impact of inulin on gut colonization with antibiotic-resistant pathogens; and (2A/exploratory) the impact of inulin on ICU-acquired antibiotic-resistant infections.

DETAILED DESCRIPTION:
The proposed trial hypothesizes that inulin maintains short-chain fatty acid (SCFA)-producing colonic anaerobes and that these bacteria are protective against multi-drug resistant organism (MDRO) colonization and subsequent MDR infection. Inulin, a vegetable-derived non-digestible polysaccharide is well established as the key nutrient source for SCFA-producing bacteria. Previous human studies have shown that (1) inulin increases levels of SCFA producers and SCFAs and (2) that this increase correlates with improved colonic mucosal integrity and resistance to MDR pathogens. In animal studies, inulin improves survival after pathogen challenge or injection with lipopolysaccharide. The overall aim of this clinical trial is to determine whether inulin improves gut colonization resistance against antibiotic-resistant pathogens and therefore prevents antibiotic-resistant infections in the setting of critical illness. To accomplish this, 90 critically ill adults who are receiving broad-spectrum antibiotics will be blindly randomized 1:1:1 to receive placebo, inulin 8 g twice daily, or inulin 16 g twice daily for a minimum of 7 days, with bedside follow-up extending to 30 days or hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized in an eligible medical ICU
2. Age ≥ 18 years old at the time of hospitalization
3. With sepsis as defined by the Sepsis-3 (2016) consensus as a known or suspected infection with a sequential organ failure assessment (SOFA) score of ≥2 points above baseline
4. Received broad-spectrum antibiotics within the last 24 hours or ordered and pending administration
5. Able to complete enrollment within 4 hours of ICU admission for administration of the intervention within 6 hours of ICU admission

Exclusion Criteria:

1. Inability to receive oral or enteric fluids
2. Inulin allergy
3. Hyponatremia (serum sodium ≤128 mEq/L)
4. Immunosuppression, defined as history of solid organ transplant or as receipt of ablative chemotherapy, steroids at the equivalent of ≥5 mg/day prednisone, antimetabolites, anti-tumor necrosis factor (TNF) α agents, calcineurin inhibitors, or mycophenolate
5. Surgery involving the intestinal lumen within 30 days or known intestinal strictures
6. Do Not Resuscitate (DNR) or Do Not Intubate (DNI) status, or "no escalation of care" orders
7. Lack capacity for consent and no appropriate Legally Authorized Representative (LAR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Freedberg, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park H, Abrams JA, Uhlemann AC, Freedberg DE. Gut Colonization With Vancomycin-Resistant Enterococcus Shapes the Gut Microbiome in the Intensive Care Unit. J Infect Dis. 2025 Sep 15;232(3):669-678. doi: 10.1093/infdis/jiaf194. PMID 40237647
- [Derived] Park H, Lynch E, Tillman A, Lewis K, Jin Z, Uhlemann AC, Abrams JA, Freedberg DE. A phase 2 randomized, placebo-controlled trial of inulin for the prevention of gut pathogen colonization and infection among patients admitted to the intensive care unit for sepsis. Crit Care. 2025 Jan 13;29(1):21. doi: 10.1186/s13054-024-05232-3. PMID 39806400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Started | 30 | 33 | 31
Completed | 30 | 30 | 30
Not Completed | 0 | 3 | 1
Not completed — Death | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [55 to 71] | 62 [44 to 69] | 65 [40 to 76] | 62 [46 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 13 | 40
  Male | 17 | 16 | 17 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 13 | 35
  Not Hispanic or Latino | 19 | 19 | 17 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 12 | 13 | 35
  Black | 5 | 7 | 7 | 19
  Other | 15 | 11 | 10 | 36
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Within-individual Change in SCFA Producer Level
Description: Relative abundance (i.e., proportion) of SCFA producing bacteria within each treatment group, will be assessed via 16S sequencing of rectal swabs. Modified intent-to-treat, comparing baseline vs Day 3 levels of SCFAs among those who receive one or more doses of the intervention and complete both assessments.
Time Frame: Baseline and Day 3
Measure: Median (Inter-Quartile Range); unit: percentage of SCFA producers
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
percentage of SCFA producers | -0.0 [-7.9 to 7.4] | -1.8 [-8.9 to 3.7] | 1.1 [-12 to 11]

2. Secondary Outcome: Multidrug Resistant Organism (MDRO)-Gram Negative Bacteria (GNB) Colonization Status
Description: Proportion of patients who are MDRO-GNB colonized within each treatment group, with MDRO-GNB colonization status classified categorically based on the presence or absence of methicillin-resistant Staphylococcus aureus (MRSA) or Gram negative bacteria (GNB) with third-generation cephalosporins non-susceptibility
Time Frame: Day 0 and at last sample collected, up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Day 0 | 6 | 4 | 3
  Last Sample Collected, Up to Day 30 | 3 | 4 | 3

3. Other Pre Specified Outcome: Fecal Short Chain Fatty Acid (SCFA) Levels
Description: The SCFAs butyrate, acetate, and propionate will be measured from whole stools on a 6490 triple quadrupole mass spectrometer and compared between intervention groups using the first stool sample produced after the Day 3 assessment. Patients who fail to produce a stool from Day 3 to 7 will be excluded from this analysis.
Time Frame: Days 3 and 7
Measure: Median (Inter-Quartile Range); unit: mMol
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
mMol
  Day 3 | 0 [0 to 0.18] | 0.11 [0 to 0.66] | 0 [0 to 0.46]
  Day 7 | 0 [0 to 0.06] | 0.29 [0 to 0.63] | 0 [0 to 0.19]

4. Other Pre Specified Outcome: ICU Length of Stay (LOS)
Description: compared between groups, after adjusting for death as a competing risk
Time Frame: through ICU Day 30
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
days | 9.5 [6 to 20] | 10.5 [6 to 23] | 9 [6 to 17]

5. Other Pre Specified Outcome: Multidrug Resistant (MDR) Infections
Description: proportion of patients with culture-proven infections within each treatment group, with culture-proven infections defined as those that have (1) an organism meeting MDRO criteria from a clinical culture, (2) signs and symptoms of infection by Centers for Disease Control (CDC)/National Health and Safety Network (NHSN) guideline definitions, and (3) receive appropriate antibiotics from the treating team
Time Frame: through 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
Participants | 15 | 9 | 12

6. Other Pre Specified Outcome: Mortality
Description: Death data will be extracted from the hospital electronic medical record (EMR) which immediately captures in-hospital death and receives monthly mortality updates from the National social security death index.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
Participants | 7 | 7 | 9

7. Secondary Outcome: Vancomycin-resistant Enterococcus (VRE) Colonization Status
Description: Proportion of patients who are VRE colonized within each treatment group, with VRE colonization status classified categorically based on the presence or absence of vancomycin-resistant Enterococcus (VRE)
Time Frame: Day 0 and at last sample collected, up to Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Day 0 | 8 | 6 | 4
  Last Sample Collected, Up to Day 30 | 11 | 13 | 6

ADVERSE EVENTS:
Time Frame: Up to Day 90
Description: Due to the severity of illness in this population (ICU patients with sepsis), only pre-specified adverse events of interest and unanticipated problems that meet the definition of a serious adverse event were collected.
Arm/Group | Placebo | Inulin 16 g/Day | Inulin 32 g/Day
All-Cause Mortality (participants affected / at risk) | 7/30 | 7/30 | 9/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 15/30 | 11/30 | 15/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Inulin 16 g/Day (N=30) | Inulin 32 g/Day (N=30)
Bloating (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 12 | 11 | 15
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Culture Proven Infection (Infections and infestations) | 15 | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03865706/Prot_SAP_001.pdf